CLINICAL TRIAL: NCT05126524
Title: Loco-regional Anaesthesia in Video or Robot-assisted Thoracic Pulmonary Surgery
Acronym: ARTIST
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: NR-2021-01
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Surgical Procedures
Keywords: Loco-regional Anaesthesia; Video or Robot-assisted Thoracic Pulmonary Surgery; ARTIST; SFAR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Loco-regional Anaesthesia in Video or Robot-assisted Thoracic Pulmonary Surgery: Patients with loco-regional Anaesthesia in Video or Robot-assisted Thoracic Pulmonary Surgery are eligible for this study
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — Observational study, no intervention performed

SUMMARY:
Currently, there is no data on the part and type of Loco-regional Anaesthesia used for Video or Robot-assisted Thoracic Pulmonary Surgery.

The aim of this epidemiological study is to identify, 6 months after the publication of the SFAR / SFCTCV 2019 recommendations, the proportion and type of Loco-regional Anaesthesia used in Video or Robot-assisted Thoracic Pulmonary Surgery within French teams.

DETAILED DESCRIPTION:
Currently, there is no data on the part and type of Loco-regional Anaesthesia used for Video or Robot-assisted Thoracic Pulmonary Surgery. The experience and habits of each team taking charge of the perioperative period seem to be the determining factors for the achievement of one type of Loco-regional Anaesthesia over another.

The aim of this epidemiological study is to identify, 6 months after the publication of the SFAR / SFCTCV 2019 recommendations, the proportion and type of Loco-regional Anaesthesia used in Video or Robot-assisted Thoracic Pulmonary Surgery within French teams.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18years and over
* Wedge surgery or lobectomy planned with Video or Robot-assisted surgery.
* non-opposition of the patient to participating in the research

Exclusion Criteria:

* Patient's refusal to use his data for research
* Emergency surgery
* Surgery with planned thoracotomy
* Contraindications to performing locoregional anesthesia
* Individual deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with planned wedge surgery or lobectomy with Video or Robot assisted surgery
Sampling Method: Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
to assess the incidence of locoregional anesthesia in video or robot-assisted thoracic pulmonary surgery | At least, 6 months after the publication of the SFAR / SFCTCV 2019 recommendations concerning this topic
  Information concerning locoregional anesthesia in video or robot-assisted thoracic are recorder in the CRF

SECONDARY OUTCOMES:
Epidemiology of anaesthesia management during Video or Robot-assisted Thoracic Pulmonary Surgery | At least, 6 months after the publication of the SFAR / SFCTCV 2019 recommendations concerning this topic
  Information concerning locoregional anesthesia in video or robot-assisted thoracic are recorder in the CRF
Epidemiology of perioperative morbidity and mortality | At least, 6 months after the publication of the SFAR / SFCTCV 2019 recommendations concerning this topic
  nformation concerning lmorbidity and mortality are recorder in the CRF

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire LE GAC, MD, Study Chair — CHU de Rennes, Hôpital de Pontchaillou
Locations (26):
- France (26):
  - CHU d'Angers, Angers
  - Hôpital Privé d'Antony, Antony
  - Clinique de l'Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - centre de Lutte Contre le Cancer Jean Perrin, Clermont-Ferrand
  - Chu Dijon, Dijon
  - CHU de Grenoble, La Tronche
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - CHRU de Lille _Clinique Cardiothoracique et Vasculaire, Lille
  - CHU Limoges, Limoges
  - Centre Leon Bérard, Lyon
  - Hôpital Nord Marseille, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHRU de Nancy, Nancy
  - CHU Nantes - Réa CTCV de l'HGR, Nantes
  - CHR d'ORLEANS, Orléans
  - Institut Mutualist Montsouris - Paris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat, Paris
  - Hôpital TENON, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Privé Claude Galien, Quincy-sous-Sénart
  - CHU de Rennes, Hôpital de Pontchaillou, Rennes
  - Polyclinique Saint Laurent, Rennes
  - CHU Charles Nicolle, Rouen
  - Centre Hospitalier de Toulon, Toulon
  - HIA Sainte-Anne - Toulon, Toulon